CLINICAL TRIAL: NCT02783209
Title: Effect on the Vitreous of the Not Complicated Surgery of the Cataract to the Emmetropic Patient
Acronym: VITRECAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Major difficulties of patient inclusions
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FME_2014_5
Record Dates: First submitted 2016-05-12; First posted 2016-05-26 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Cataract; Vitreous Detachment
MeSH Terms: conditions — Cataract; Vitreous Detachment | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cataract surgery (Other): Patient acts as his own control
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Procedure: Cataract surgery

SUMMARY:
This study evaluates the association between surgery of the cataract and posterior vitreous detachment, in the emmetropic patient, by comparing eyes operated with eyes not operated in the same group of patients

ELIGIBILITY:
Inclusion Criteria:

* Adult emmetropic patient
* Without complete posterior vitreus detachment in both eyes before having surgery.

Exclusion Criteria:

* Diabetic retinopathy
* Ophthalmological treatment in progress
* History of ophthalmological surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Occurence of vitreous detachment in the operated eye | 3 months after the cataract surgery

CONTACTS AND LOCATIONS:
Locations (1):
- URC Fondation Ophtalmologique A de Rothschild, Paris, France